CLINICAL TRIAL: NCT02452372
Title: A Phase 1, Single-ascending Dose, Multiple-ascending Dose, and Multi-dose Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of Subcutaneously Administered ALN AS1 in Patients With Acute Intermittent Porphyria (AIP)
Brief Title: A Phase 1 Study of Givosiran (ALN-AS1) in Patients With Acute Intermittent Porphyria (AIP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALN-AS1-001
Record Dates: First submitted 2015-05-19; First posted 2015-05-22 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Acute Intermittent Porphyria
Keywords: RNAi therapeutic; Porphyria; AIP
MeSH Terms: conditions — Porphyria, Acute Intermittent; Porphyrias | interventions — givosiran

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- givosiran (ALN-AS1) (Active Comparator)
  Interventions: Drug: givosiran (ALN-AS1)
- Sterile Normal Saline (0.9% NaCl) (Placebo Comparator)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: givosiran (ALN-AS1) — Single or multiple doses of ALN-AS1 by subcutaneous (sc) injection
  Arms: givosiran (ALN-AS1)
Drug: Sterile Normal Saline (0.9% NaCl) — calculated volume to match active comparator
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of givosiran (ALN-AS1) in AIP patients as well as to characterize pharmacokinetics (PK) and pharmacodynamics (PD) of ALN-AS1 in AIP patients.

ELIGIBILITY:
Parts A and B

Inclusion Criteria:

* Diagnosis of AIP
* Urine PBG at Screening indicating patient is a high excreter
* No clinically significant health concerns
* Women of child bearing potential must have a negative pregnancy test, not be nursing, and use effective contraception
* Willing to provide written informed consent and willing to comply with study requirements.

Exclusion Criteria:

* Porphyria attack within 6 months of screening
* Started a new prescription medication within 3 months of screening
* Clinically significant abnormal laboratory results
* Received an investigational agent within 90 days before the first dose of study drug or are in follow-up of another clinical study
* History of multiple drug allergies or intolerance to subcutaneous injection

Part C

Inclusion Criteria:

* Diagnosis of AIP
* Patient experienced a porphyria attack or was taking medication to prevent attacks recently
* No clinically significant health concerns
* Women of child bearing potential must have a negative pregnancy test, not be nursing, and use effective contraception
* Willing to provide written informed consent and willing to comply with study requirements.

Exclusion Criteria:

* Stared a new prescription medication within 3 months of screening
* Clinically significant abnormal laboratory results
* Received an investigational agent within 90 days before the first dose of study drug or are in follow-up of another clinical study
* History of multiple drug allergies or intolerance to subcutaneous injection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
The safety of givosiran evaluated by the proportion of subjects experiencing adverse events (AEs), serious adverse events (SAEs), and AEs leading to study drug discontinuation | Part A (SAD phase): through day 42; Part B (MAD) phase: through Day 70; Part C (MD) phase: through Day 168

SECONDARY OUTCOMES:
Profile of Pharmacokinetics (PK) of givosiran | Part A (SAD) phase: predose - 42 days post-dose; Part B (MAD) phase: predose - 70 days post-dose; Part C (MD) phase: predose - 168 days post-dose
  Cmax
Profile of Pharmacokinetics (PK) of givosiran | Part A (SAD) phase: predose - 42 days post-dose; Part B (MAD) phase: predose - 70 days post-dose; Part C (MD) phase: predose - 168 days post-dose
  tmax
Profile of Pharmacokinetics (PK) of givosiran | Part A (SAD) phase: predose - 42 days post-dose; Part B (MAD) phase: predose - 70 days post-dose; Part C (MD) phase: predose - 168 days post-dose
  AUC
Profile of Pharmacokinetics (PK) of givosiran | Part A (SAD) phase: predose - 42 days post-dose; Part B (MAD) phase: predose - 70 days post-dose; Part C (MD) phase: predose - 168 days post-dose
  t1/2
The change in delta-aminolevulinic acid (ALA) from baseline | Part A (SAD) phase: screening - 42 days post-dose; Part B (MAD) phase: screening - 70 days post-dose; Part C (MD) phase: screening - 168 days post-dose
The change in Porphobilinogen (PBG) from baseline | Part A (SAD) phase: screening - 42 days post-dose; Part B (MAD) phase: screening - 70 days post-dose; Part C (MD) phase: screening - 168 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Amy Simon, MD, Study Director — Alnylam Pharmaceuticals
Locations (6):
- United States (4):
  - Clinical Trial Site, Birmingham, Alabama
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Galveston, Texas
- Clinical Trial Site, Stockholm, Sweden
- Clinical Trial Site, London, United Kingdom

REFERENCES:
- [Derived] Sardh E, Balwani M, Rees DC, Anderson KE, Jia G, Sweetser MT, Wang B. Long-term follow-up of givosiran treatment in patients with acute intermittent porphyria from a phase 1/2, 48-month open-label extension study. Orphanet J Rare Dis. 2024 Oct 3;19(1):365. doi: 10.1186/s13023-024-03284-w. PMID 39363243
- [Derived] Sardh E, Harper P, Balwani M, Stein P, Rees D, Bissell DM, Desnick R, Parker C, Phillips J, Bonkovsky HL, Vassiliou D, Penz C, Chan-Daniels A, He Q, Querbes W, Fitzgerald K, Kim JB, Garg P, Vaishnaw A, Simon AR, Anderson KE. Phase 1 Trial of an RNA Interference Therapy for Acute Intermittent Porphyria. N Engl J Med. 2019 Feb 7;380(6):549-558. doi: 10.1056/NEJMoa1807838. PMID 30726693